CLINICAL TRIAL: NCT03186612
Title: Effects of a Game-based Virtual Reality Video Capture Training Program Plus Occupational Therapy on Manual Dexterity in Patients With Multiple Sclerosis: a Randomizaed Controlled Trial
Brief Title: Virtual Reality and Manual Dexterity in in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversidadRJC
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis; Physical Activity; Upper Limb; Virtual Reality; Dexterity
Keywords: Video games; Virtual reality; Occupational therapy, Manual dexterity; Multiple sclerosis.
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: It will be conducted a blinded randomized controlled trial (RCT). Non-probabilistic sampling of consecutive cases will be used.
Who Masked: Outcomes Assessor
Masking Description: All assessments were conducted by masked evaluators. They were not related to the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT intervention (Active Comparator): Conventional occupational therapy (OT) treatment will consist of 20 sessions in total, during which subjects will perform activities for training manipulative and functional dexterity of the upper limb aimed at activities of daily living. These will be distributed in two OT sessions per week, each lasting 30 minutes.
  Interventions: Behavioral: OT+VR intervention with videogames for the upper limb (dexterity)
- OT+VR intervention (Experimental): The intervention applied to the experimental group will consist of 20 sessions of conventional OT distributed in two sessions per week, each lasting 30 minutes. Additionally, they will receive 20 treatment sessions lasting 20 minutes, twice weekly of virtual reality (VR) via the online and free website motiongamingconsole.com, during which they will performe exercises with video capture of the upper limb movements via the performance of functional and manual dexterity activities based on the following games: Flip Out, Air Hockey, Particlesículas, Dunkit, Cuenta PecesCounting fishes and Robo Maro. All the interventions will consider the level of fatigue experimented by the patient by featuring a progressive increase of the treatment times according to the same.
  Interventions: Behavioral: OT+VR intervention with videogames for the upper limb (dexterity)

INTERVENTIONS:
Behavioral: OT+VR intervention with videogames for the upper limb (dexterity) — Patients will performe exercises with video capture of the upper limb movements via the performance of functional and manual dexterity activities based on the following games: Flip Out, Air Hockey, Particlesículas, Dunkit, Cuenta PecesCounting fishes and Robo Maro.

SUMMARY:
Introduction. Multiple sclerosis (MS) is the most common neurological disease causing disability in young adults. Neurorehabilitation is a fundamental aspect in the treatment approach for MS, in which new technologies have gained popularity, especially the use of virtual reality (VR), thanks to the therapeutic possibilities offered for patients with MS presenting cognitive, sensitive and motor dysfunctions.

Aim. To analyze and compare an occupational therapy intervention (OT) compared with OT + VR (OT+VR) on the manual dexterity of patients with MS.

Material and methods. 26 patients will be recruited. The control group (n=8) will recieve 20 conventional OT sessions distributed in two sessions per week. The experimental group OT+VR (n=8) will recieve 20 sessions of VR interventions, twice weekly and lasting 30 minutes, consisting of VR games accessed via the online webpage motiongamingconsole.com, including Flip Out, Air Hockey, Partículas, Dunkit, Cuenta peces and Robo Maro, in addition to the conventional OT sessions. Pre and post-intervention assessments will be based on the Purdue Pegboard Test, the Jebsen Taylor Hand Function Test and the Grooved Pegboard Test.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating illness of the central nervous system (CNS) of unknown etiology and a multifactorial origin. Currently, MS represents the most common neurological illness that causes disability among young adults in Europe and North America.

The symptoms depend on the areas of the CNS that are injured, with considerable clinical variability between patients, depending on the level of severity and the duration of the disease. Among the most common symptoms, patients exhibit fatigue, visual disorders, problems affecting balance and coordination, sensitivity disorders, spasticity, cognitive and emotional disorders, speech disorders, problems affecting the bladder and intestines, as well as sexual related dysfunction.

Different disease courses exist for MS, according to the appearance of symptoms, such as relapsing-remitting MS, primary progressive MS, secondary-progressive MS and progressive-recurrent MS. Relapsing-remitting MS is the most common form of MS.

The symptoms appear in the form of relapses, which are of a variable duration and which vary from one episode to the other, according to the affected area in the CNS. After the flare-ups, symptoms subside and usually disappear completely, although there may be neurological aftereffects. In primary-progressive MS, a progressive clinical deterioration occurs, without relapses, from the onset of the illness. This type of MS is suffered by 12% of people with MS. In secondary-progressive MS, patients initially present a relapsing-remitting course, however, over time, they develop a progressive clinical deterioration without experiencing distinctive relapses. Progressive-recurrent MS, is the least common type of illness.

Two fundamental and complementary aspects exist in the treatment of MS: pharmacological and rehabilitation treatments. Over recent years, a substantial change has occurred in the approach to MS, thanks to the appearance of new drugs aimed at modifying the progression of the disease. However, these drugs would be more effective if they were complemented by a good rehabilitation program. With regards rehabilitation, a symptomatic treatment of MS is performed in order to improve the quality of life and functional independence, with the main therapeutic demands being the alterations of postural control and the performance of activities of daily living. Occupational therapy (OT) assesses the capacities and physical, psychological, sensory and social problems of the individual with MS, in order to enable the person to achieve the greatest possible level of independence in their daily living and/or to facilitate the adaptation to their disability. At times, rehabilitation treatments for patients with MS can be very lengthy and systematic, leading to patients that lose motivation and compliance. As a result, in recent years, new intervention strategies have been introduced, such as virtual reality (VR), thanks to VR motion capture technology without the need of using any device or controller. Here, patient motivation is promoted via novel approaches based on practicing functional tasks in virtual surroundings, which provide feedback to the patient concerning results, and are based on the repetition of activities of daily living (ADLs). The development of these technologies has provided rehabilitation professionals with the ability to expand the care of patients with MS as a complement to their rehabilitation program, achieving a higher treatment intensity at a sustainable cost. However, there are few studies on the effects that VR has on the manual dexterity of patients with MS.

Therefore, the objective of the present study was to analyze the effects of an OT intervention combined with VR on manual skills, compared with conventional OT approaches in people with MS.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of MS according to the McDonald criteria with over two years evolution;
* a score of between 3.5 (moderate incapacity, although totally ambulant and able to be self-sufficient and active during 12 hours of a day) and six (requires constant help, either unilateral or intermittently with a walking stick or crutches, in order to walk approximately 100 meters with, or without, a rest) on the Kurtzke Expanded Disability Status Score (EDSS) with;
* stable medical treatment during, at least the six months prior to the intervention;
* muscle tone in the upper limbs not greater than two points on the modified Ashworth Scale (moderate hypertonia, increased muscle tone through most of the range of movement, but affected part easily moved);
* as well as a score of four points or less in the "Pyramidal Function" section of the EDSS functional scale;
* absence of cognitive decline; with the ability to understand instructions and obtaining a score of 24 or more in the Minimental Test;
* as well as a score of two points or less in the "Mental Functions" section of the EDSS.

Exclusion Criteria:

* the diagnosis of another neurological illness or musculoskeletal alteration different to MS;
* the diagnosis of a cardiovascular, respiratory or metabolic illness, or other conditions which may interfere with the study;
* suffering a flare-up or hospitalization in the last three months prior to commencement of the assessment protocol, or during the process of the therapeutic intervention;
* receiving a cycle of steroids, either intravenously or oral, six months prior to the commencement of the assessment protocol and within the study period of intervention;
* receiving treatment with botulinum toxin in the six months prior to the beginning of the study; or the presence of visual disorders non-corrected by optical devices.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-12-02 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Manual dexterity, gross dexterity and coordination | 2 mothns and 15 days between assessments. The "change" that it is being assessed is fine manual dexterity
  It will be used Purdue Pegboard Test (PPT) for the assessment gross dexterity and coordination. This test assesses the speed and motor dexterity of each hand and the manual dexterity using both hands at the same time. The PPT consists of a board with two columns with 25 holes each and a specific number of pins, washers and collars placed in four containers across the top of the board. The test consists of inserting as many pins as possible in three distinct phases, with a time limit of 30 seconds for each part. First, the test is performed with the dominant hand, then with the non-dominant hand and then with both hands at the same time. The number of pins inserted is recorded.
Hand´s functional capacity | 2 mothns and 15 days between assessments. The "change" that it is being assessed is hand's functional status
  The Jebsen Taylor Hand Function Test (JTT) will be used to determine the hand's functional capacity. This test is timed and divided in seven parts. The seven subtests are: writing, page turning, picking up small common objects, simulated feeding, stacking checkers, moving large light objects and moving large heavy objects.
  All the subtests are performed with the dominant hand first, followed by the dominant hand. The time the subject takes to perform each subtest is recorded.
Manipulative dexterity | 2 mothns and 15 days between assessments. The "change" that it is being assessed is manipulative dexterity
  The Grooved Pegboard Test (GPT) is a test that evaluates manipulative dexterity. This test is performed with the dominant hand and consists of inserting pegs in the slots of a board which are placed at different angles. The score is the time in seconds required for inserting all the pegs.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cano de la Cuerda, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Roberto Cano de la Cuerda, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortiz-Gutiérrez R, Galán del Río F, Cano de la Cuerda R, Alguacil Diego IM, Arroyo-González R, Miangolarra-Page JC.A telerehabilitation program by virtual reality-video games improves balance and postural control in multiple sclerosis patients. NeuroRehabilitation. 2013; 33(4):545-54. Ortiz-Gutiérrez R, Cano-de la Cuerda R, Galán-del Río F, Alguacil-Diego IM, Palacios-Ceña D, Miangolarra-Page JC. A telerehabilitation program improves postural control in multiple sclerosis patients. A Spanish preliminary study. Int J Environ Res Public Health 2013;10(11):5697-710 Palacios-Ceña D, Ortiz-Gutierrez R, Buesa-Estellez A, Galán-del-Río F, Cachón- Pérez JM, Martinez-Piédrola R, Velarde-García JF, Cano-de-la-Cuerda R. Multiple sclerosis patients' experiences in relation to the impact of the kinect virtual home- exercise programme: a qualitative study. Eu J Phys Rehabil Med 2016;52(3):347-55. Shin JH, Kim MY, Lee JY, Jeon YL, Kim S, Lee S, Seo B, Choi Y. Effects of virtual reality-based rehabilitation on distal upper extremity function and health-related quality of life: a single-blinded, randomized controlled trial. J Neuroeng Rehabil. 2016; 13:17.